CLINICAL TRIAL: NCT00466037
Title: Vaccination Against Influenza in Rheumatoid Arthritis Patients: The Effect of Rituximab on the Humoral Response
Brief Title: The Effect of Rituximab on the Humoral Response to Influenza Vaccine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-05-OE-204-CTIL
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid; rituximab; influenza
MeSH Terms: conditions — Arthritis, Rheumatoid; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Influenza vaccine

SUMMARY:
Rituximab is a genetically engineered chimeric anti-CD20 monoclonal antibody that selectively targets CD20+ B cells and induces a transient depletion of the CD20+ mature B cell subpopulation.The objective of our study was to assess the effect of rituximab on the efficacy and safety of influenza virus vaccine in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The study population comprised RA patients treated with conventional disease modifying drugs with or without rituximab. Split-virion inactivated vaccine containing 15 mcg hemagglutinin/dose of B/Shanghai/361/02 (SHAN), A/New Caledonia A/New Caledonia/ 20/99 (NC) (H1N1) and A/California/7/04 (CAL) (H3N2) was used. Disease activity was assessed by number of tender and swollen joints, morning stiffness duration, and evaluation of pain on the day of vaccination and 4 weeks later. CD20 positive cell levels were assessed in rituximab treated patients. Hemagglutination inhibition (HI) antibodies were tested and response was defined as >4-fold rise 4 weeks post vaccination or seroconversion in patients with a non-protective baseline level of antibodies (<1/40). Geometric mean titers (GMT) were calculated in all subjects.

Results: The participants were divided into 3 groups: RA (n=29, aged 64±12 years), rituximab-treated RA (n=14, aged 53±15 years) and healthy controls (n=21, aged 58±15 years). All baseline protective levels of HI antibodies and GMT were similar. Four weeks after vaccination, there was a significant increase in GMT for NC and California antigens in all subjects, but not for the Shanghai antigen in the rituximab group. Similarly, the percentage of responders was low for Shanghai and NC, but significantly lowers in rituximab treated patients for the California antigen compared with the other groups. Parameters of disease activity remained unchanged.

Conclusion: Influenza virus vaccine generated a humoral response in all RA study patients and controls. Although the response was significantly lower among rituximab-treated patients,

ELIGIBILITY:
Inclusion Criteria:

* Patients with Rheumatoid Arthritis
* Age-18-85
* Treatment with Rituximab and other Disease modifying drugs

Exclusion Criteria:

* Treatment with anti TNF alpha
* Allergy to eggs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2005-09; Study Completion 2006-02

PRIMARY OUTCOMES:
Efficacy of vaccination against influenza

SECONDARY OUTCOMES:
Safety of vaccination against influenza in Rheumatoid Arthritis patients

CONTACTS AND LOCATIONS:
Overall Officials: Ori Elkayam, M.D, Principal Investigator — Tel Aviv Medical Center